CLINICAL TRIAL: NCT01949753
Title: Influence of Pregnenolone on Distress and Autonomic Parameters During Cognitive-behavioral Exposure Therapy in Patients With Obsessive-compulsive Disorder
Brief Title: Influence of Pregnenolone on Exposure Therapy in Obsessive-compulsive Disorder
Acronym: P-EX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PV4398
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Obsessive-compulsive Disorder (OCD)
Keywords: Obsessive-compulsive disorder (OCD); Exposure therapy; Extinction learning; Pregnenolone
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplement Pregnenolone (Experimental): Exposure therapy, exposure with response prevention and pharmacological facilitation (nutritional supplement pregnenolone), orally two hours before exposure therapy.
  Interventions: Behavioral: Exposure therapy with pharmacological facilitation
- Placebo (Placebo Comparator): Exposure therapy, exposure with response prevention without pharmacological facilitation (Placebo), orally two hours before exposure therapy.
  Interventions: Behavioral: Exposure therapy

INTERVENTIONS:
Behavioral: Exposure therapy with pharmacological facilitation — Exposure with response prevention and pharmacological facilitation
  Arms: Nutritional supplement Pregnenolone
Behavioral: Exposure therapy — Exposure with response prevention without pharmacological facilitation
  Arms: Placebo

SUMMARY:
Characterization of the influence of pregnenolone vs. placebo on subjective distress and autonomic functioning during cognitive-behavioral exposure therapy in patients with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
Main out-come parameters:

Inter-session habituation as per SUD (100 mm VAS), Y-BOCS

Secondary out-come parameter:

HF/LF of HRV, Salivary epinephrine

ELIGIBILITY:
Inclusion Criteria:

-OCD according to DSM-IV criteria.

Exclusion Criteria:

* Acute suicidality
* psychotic disorders,
* bipolar disorder
* substance dependency
* organic brain disorder
* pregnancy
* lactation
* tuberculosis
* gastric/duodenal ulcer
* diabetes mellitus
* acute inflammation
* autoimmune disorders
* arterial hypertension
* therapy with glucocorticoids (up to 4 weeks ago)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Subjective units of distress (SUD) | During exposure therapy

SECONDARY OUTCOMES:
Low/high frequency index of heart rate variability (L/HFI) | During exposure therapy

OTHER OUTCOMES:
Salivary cortisol, noradrenaline, pregnenolone; heart rate, blood pressure | During exposure therapy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kellner, MD, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Hospital Hamburg-Eppendorf, Hamburg, Germany